CLINICAL TRIAL: NCT03481179
Title: Efficacy of High Frequency Repetitive Transcranial Magnetic Stimulation Associated With Physical Therapy to Reduce Upper Limb Spasticity in Post Stroke Patients: Double Blinded, Randomized and Controlled Clinical
Brief Title: Repetitive Transcranial Magnetic Stimulation Associated With Physical Therapy to Reduce Upper Limb Spasticity in Post Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Kátia Monte-Silva, principal investigator, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Stroke_High_rTMS
Record Dates: First submitted 2018-02-01; First posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Chronic Stroke
Keywords: Repetitive transcranial magnetic stimulation, Physiotherapy, Stroke, Spasticity
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: hf rTMS and Physical therapy (Experimental): High frequency TMS will be applied with an eight shaped coil angled at 45 degrees from the sagittal axis and positioned at the C3 or C4 in accordance with the international 10-20 marking system (JASPER, 1958), which corresponds to the right or left primary motor cortex (M1) injured. Forty stimulus trains will be provide at 10Hz over the injured hemisphere, at 10 Hz for five seconds each. The interval between the trains will be 25 seconds, totaling 2000 pulses for approximately 20 minutes, with 120% of resting motor threshold (RMT). After TMS, patients will be submitted to 50 minutes of physical therapy protocol.
  Interventions: Device: TMS; Other: Physical therapy
- Control: Sham hf rTMS and Physical theraphy (Sham Comparator): In this group, the volunteer will start with sham TMS, will be the same parameters was used in experimental group, however, it will be performed using two coils, one connected to the magnetic stimulator, away from the patient's scalp and another uncoupled from the stimulator and positioned in the same way as in real stimulation. After, the volunteer will be submitted to 50 minutes of physical therapy protocol.
  Interventions: Device: TMS; Other: Physical therapy

INTERVENTIONS:
Device: TMS — Repetitive TMS involves application of electric currents in the patient's cortex by a magnetic field applied to the scalp of the patient through an eight-coil connected to a magnetic stimulator (MagStim Rapid² magnetic stimulator-UK). In a small percentage of patients, it may cause some discomfort with a mild headache sensation or nausea. Depending on the parameters, rTMS can increase or decrease corticomotor excitability and by the connection of the motor cortex with the thalamus, influencing spasticity inhibition. The patients will respond to an adverse effects questionnaire and will report the perception of real or sham stimulation.
  Other Names: non invasive brain stimulation, high frequency rTMS
Other: Physical therapy — The physical therapy, with an duration of 40-50 minutes, will be focused on the upper limbs and will be based on the principles of neuroplasticity (repetition, intensity, specificity, among others (KLEIM & JONES, 2008), with a protocol that will cover different exercises and degrees of difficulty, which will be chosen according to the need and capacity of each patient

SUMMARY:
In this study, it is being investigated if the association between high frequency repetitive transcranial magnetic stimulation associated with motor physical therapy reduces spasticity, increases upper limb motor function, and quality of life of post-chronic stroke patients than motor physical therapy alone. For this purpose, patients included will be submitted to ten sessions with active or sham hf-rTMS followed by a protocol of physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 to 75 years;
* Both sexes;
* With diagnosis of ischemic or hemorrhagic stroke proven by means of computed tomography or magnetic resonance imaging;
* Spasticity grade will be assessed using the Ashworth modified scale (BOHANNON & SMITH, 1987), with score +1, 2 or 3 for the wrist flexors of the affected upper limb;
* With absence of cognitive deficit verified by the Folstein Mini Mental State Examination (score ≥ 20) modified for the Brazilian population (BRUCKI et al., 2003)

Exclusion Criteria:

* Contraindications to and EMT (ROSSINI et al., 2015)
* Clinical evidence of multiple brain lesions
* Trauma-orthopedic injury that limits the range of motion of the upper limb
* Presence of visual and / or communication deficit
* Involvement of other interventions focused on reducing spasticity
* Modification of medications in the last 30 days.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Spasticity | before 10 sessions, before and after each session (every day), after 10 daily sessions and after 30 days
  Change from degree of Spasticity: ordinal variable measured through the Ashworth Modified Scale, expressed as scores graded from +1 to 3. The EMA is a qualitative instrument with ordinal measures that scores the degree of spasticity presented by the resting muscle from zero to four, in increasing order of intensity.

SECONDARY OUTCOMES:
Cortical excitability | before and after 10 daily sessions and after 30 days
  Expressed as percent motor resting threshold and numerical values of motor evoked potential. The motor evoked potential (MEP) will be provided by twenty unconditioned stimuli (120% of motor resting threshould).
Variation of the median nerve Hmax / Mmax ratio | before and after 10 sessions and after 30 days
  The reflex H is an estimate of the excitability of the alpha motoneuron when there is a pre-synaptic inhibition (PALIERI, R.M et al., 2004). The variation of the H-reflex amplitude will evaluate the spinal cord excitability variation.
Sensory-motor function of the upper limb | before and after 10 daily sessions and after 30 days
  This consists of a quantitative scale developed to measure the recovery of the motor function of stroke patients.Measured through the Fugl-Meyer Rating Scale. Expressed in values from 0 to 66;
Quality of life | before and after 10 daily sessions and after 30 days
  Expressed in numerical values for each domain, the SSQOL has 49 items distributed in 12 domains (energy, family role, language, mobility, humor, personality, self-care, social role, reasoning, upper limb function, vision and work / productivity). There are three possibilities for responses that are quantified on a five-to-one scale.
Qualitative and quantitative of moviment | before and after 10 daily sessions and after 30 days
  Motor Activity Log 30 (MAL-30) is a standardized instrument that was developed specifically to evaluate the function and use of the upper limb most affected post-stroke in the real-life environment (uncontrolled) through two scales: qualitative and quantitative. The total score is obtained by calculating the mean for each of the scales. The higher the mean obtained in the scales, the better the quality and quantity of use of the upper limb more affected in the accomplishment of the daily activities of life.
Dynamometry | before and after 10 daily sessions and after 30 days
  It consists of an objective and quantitative way of measuring muscle shape using a manual portable dynamometer. The test will be performed with the Jamar dynamometer in KGF.
Changes on Patient Global Impression of Change Scale | before and after 10 daily sessions and after 30 days
  Changes on Patient Global Impression of Change Scale - (time frame: baseline, before 6 session, after 10 sessions)
  The PGICS is a one-dimensional measure in which individuals rate their improvement associated with intervention on a scale of 7 items ranging from "1 = no change" to "7 = Much better".

CONTACTS AND LOCATIONS:
Overall Officials: Kátia Monte-Silva, PhD, Study Director — Applied Neuroscience Laboratory, Universidade Federal de Pernambuco
Locations (1):
- Applied Neuroscience Laboratory, Recife, Pernambuco, Brazil